CLINICAL TRIAL: NCT03007225
Title: Efficacy and Safety of Drug Eluting Beads TACE in Treatment of HCC in Egyptian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate professor of tropical medicine , Ain Shams university, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: treatment of HCC
Record Dates: First submitted 2016-12-24; First posted 2017-01-02 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 Drug eluting beads intervention (Active Comparator): Twenty-five patients underwent Chemoembolization with Drug eluting beads. using Drug eluting Doxorubicin hydrochloride (100-150 mg)
  Interventions: Drug: TACE with Drug Eluting Beads procedure
- group 2 Conventional TACE intervention (Active Comparator): Twenty-five patients underwent conventional Chemoembolization (cTACE) using the standard TACE technique
  Interventions: Drug: Trans-arterial chemoembolization (TACE)

INTERVENTIONS:
Drug: Trans-arterial chemoembolization (TACE) — TACE procedures were performed by experienced radiologists by fluoroscopy. The femoral artery was catheterized under local anesthesia, with a 4F catheter with Copra head configuration. Conventional angiography of the Coeliac and Hepatic arteries to delineate the feeding arteries of the tumors and to exclude portal venous shunting. Then vascular catheter was inserted super-selectively into the branch of the hepatic artery that is the main feeder of the tumor. Chemoembolization then was performed.
  Ten milliliters of Lipiodol was mixed with 100 mg of Doxorubicin hydrochloride and 5ml of Urografin emulsified to create a milky solution. The emulsion slowly was infused into the tumour Gel foam embolization was performed by cutting gel foam sheets into small pledges mannully then mixed with a contrast material and an impirical antibiotic (gentamycin 80 mg). Injection of the mixture slowly under fluoroscopy guidance till complete stasis was achieved.
  Other Names: TACE
  Arms: group 2 Conventional TACE intervention
Drug: TACE with Drug Eluting Beads procedure — The same was done as cTACE till the super selective catheterization of the feeding artery.
  Loading of the beads with Doxorubicin hydrochloride (100-150 mg) was done in vitro an hour before the beginning of catheterization. The loaded beads were then aspirated from the vial into a syringe filled with nonionic contrast medium. Once the feeding artery was identified and catheter was in placement, the loaded beads were infused slowly under fluoroscopic guidance. Two different sizes of DC beads were used, 100-300 μm and 300-500. Starting with the smaller sized beads to occlude the tumoral bed followed by the larger sized one to embolize the proximal vessels. The injection of the loaded beads was performed as selective as possible using either a4F diagnostic catheter (Cobra head catheter; Cordis, USA) or 2.7F microcatheter (Progreat; Terumo, Japan).
  Other Names: DEB-TACE
  Arms: group 1 Drug eluting beads intervention

SUMMARY:
This study aimed to to compare the conventional transarterial chemoembolization (cTACE) with chemoembolization using doxorubicin drug eluting beads (DEB-TACE) for the treatment of hepatocellular carcinoma regarding short term efficacy and safety in first 3 months after embolization

DETAILED DESCRIPTION:
This prospective case control was conducted at the Department of Tropical Medicine and HCC Clinic, Ain Shams University Hospitals (Cairo, Egypt), The patients were divided according to the line of treatment into 2 groups:

1. Group (I): Twenty-five patients underwent Chemoembolization with Drug eluting beads.
2. Group (II): Twenty-five patients underwent conventional Chemoembolization (cTACE)

The total number of procedures was 77 sessions (37 sessions of TACE with beads and 40 sessions of conventional TACE).Post-procedure follow up:

Schedule of follow up:

All included patients were checked at:

1. One week after the procedure to detect early post chemoembolization complications and Patients were subjected to Liver function tests, Kidney function tests, complete blood count and Abdominal Ultrasound.
2. One and four months after the maneuver.

Patients were subjected to the following in each visit:

1. Complete History taking
2. Thorough clinical examination
3. Laboratory Investigations including:

   1. Liver function tests
   2. Kidney function tests
   3. CBC
   4. Serum alpha-fetoprotein.
4. Triphasic pelvi-abdominal CT Follow up imaging was performed at the first and fourth months after embolization and every 3 months thereafter. Repeated embolization was scheduled "on demand" basis, if there was residual viable tumor deemed unsuitable for radiofrequency ablation or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC according to the European association of study of liver diseases
* Early stage HCC (Stage A), using the Barcelona Clinic Liver Cancer (BCLC) staging system, (single or 3 nodules < 3cm PS 0) whenever curative measures were contraindicated and BCLC stage B (intermediate HCC).
* Patent portal vein and its main branches
* Informed consent from all participants before enrollment in the study.

Exclusion Criteria:

* Patients with Child class C according to Child classification (BCLC D).
* Patients with diffuse HCC (non-measurable lesion).
* Patients with thrombosis of main portal vein or one of its main branches (BCLC C).
* Patients with extra hepatic invasion.
* patients refused to participate in the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment finished and study completed Patients collected from HCC clinic full filling the inclusion criteria,Ain Shams University hospitals
Groups:
- Chemoembolization + Drug Eluting Beads: Twenty-five patients underwent Chemoembolization with Drug eluting beads. using Drug eluting Doxorubicin hydrochloride (100-150 mg)
  TACE with Drug Eluting Beads procedure: The same was done as cTACE till the super selective catheterization of the feeding artery.
  Loading of the beads with Doxorubicin hydrochloride (100-150 mg) was done in vitro an hour before the beginning of catheterization. The loaded beads were then aspirated from the vial into a syringe filled with nonionic contrast medium. Once the feeding artery was identified and catheter was in placement, the loaded beads were infused slowly under fluoroscopic guidance. Two different sizes of DC beads were used, 100-300 μm and 300-500. Starting with the smaller sized beads to occlude the tumoral bed followed by the larger sized one to embolize the proximal vessels. The injection of the loaded beads was performed as selective as possible using either a4F diagnostic catheter or 2.7F microcatheter
- Chemoembolization + Standard TACE Technique: Twenty-five patients underwent conventional Chemoembolization (cTACE) using the standard TACE technique
  Trans-arterial chemoembolization (TACE): TACE procedures were performed by experienced radiologists by fluoroscopy. The femoral artery was catheterized under local anesthesia, with a 4F catheter . Conventional angiography of the Coeliac and Hepatic arteries to delineate the feeding arteries of the tumors and to exclude portal venous shunting. Then vascular catheter was inserted super-selectively into the branch of the hepatic artery that is the main feeder of the tumor. Chemoembolization then was performed.
  Ten milliliters of Lipiodol was mixed with 100 mg of Doxorubicin hydrochloride and 5ml of Urografin emulsified to create a milky solution.
  Gel foam embolization was performed then mixed with a contrast material and an impirical antibiotic (gentamycin 80 mg). Injection of the mixture slowly under fluoroscopy guidance till complete stasis was achieved.
Period: Overall Study
Arm/Group | Chemoembolization + Drug Eluting Beads | Chemoembolization + Standard TACE Technique
Started (Study completed) | 25 (Followed up for at least 6 months after DEB TACE) | 25 (followed up for at least 6 months after TACE)
Completed (Study completed) | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Twenty-five patients underwent Chemoembolization with Drug eluting beads. using Drug eluting Doxorubicin hydrochloride (100-150 mg)
  The procedure: The same was done as cTACE till the super selective catheterization of the feeding artery.
  Loading of the beads with Doxorubicin hydrochloride was done in vitro an hour before the beginning of catheterization. The loaded beads were then aspirated from the vial into a syringe filled with nonionic contrast medium. Once the feeding artery was identified and catheter was in placement, the loaded beads were infused slowly under fluoroscopic guidance. Two different sizes of DC beads were used, 100-300 μm and 300-500. Starting with the smaller sized beads to occlude the tumoral bed followed by the larger sized one to embolize the proximal vessels. The injection of the loaded beads was performed as selective as possible using either a4F diagnostic catheter (Cobra head catheter; Cordis, USA) or 2.7F microcatheter (Progreat; Terumo, Japan).
- Group 2: Twenty-five patients underwent conventional Chemoembolization (cTACE) using the standard TACE technique
  TACE procedures were performed by experienced radiologists by fluoroscopy. The femoral artery was catheterized under local anesthesia, with a 4F catheter with Copra head configuration. Conventional angiography to delineate the feeding arteries of the tumors and to exclude portal venous shunting. Then vascular catheter was inserted super-selectively into the branch of the hepatic artery that is the main feeder of the tumor. Chemoembolization then was performed.
  Ten milliliters of Lipiodol was mixed with 100 mg of Doxorubicin hydrochloride and 5ml of Urografin emulsified to create a milky solution. The emulsion slowly was infused into the tumour Gel foam embolization was performed and an impirical antibiotic (gentamycin 80 mg). Injection of the mixture slowly under fluoroscopy guidance till complete stasis was achieved.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (6.8) | 56 (5.5) | 56.7 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants] — 50 HCC patients entered the study collected from Our weekly HCC clinic,Ain Shams University hodpilals fullfilling the inclusion criteria and after explaining the trial to the patients and obtained informed Vincent from wash patients
  Participants
    Female | 4 | 3 | 7
    Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 25 | 25 | 50
50 patients with HCC collected from our weekly HCC clinic, Ain Shams University Hospitals [Count of Participants; unit: Participants] | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Assessment of Radiological response by modified RECIST radiological criteria after treatment (Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.")
Time Frame: 1 year
Measure: Number; unit: Participants
Groups:
- Group 1: Twenty-five patients underwent Chemoembolization with Drug eluting beads. using Drug eluting Doxorubicin hydrochloride (100-150 mg)
  TACE with Drug Eluting Beads procedure: The same was done as cTACE till the super selective catheterization of the feeding artery.
  Loading of the beads with Doxorubicin hydrochloride was done in vitro an hour before the beginning of catheterization. The loaded beads were then aspirated from the vial into a syringe filled with nonionic contrast medium. Once the feeding artery was identified and catheter was in placement, the loaded beads were infused slowly under fluoroscopic guidance. Two different sizes of DC beads were used, 100-300 μm and 300-500. Starting with the smaller sized beads to occlude the tumoral bed followed by the larger sized one to embolize the proximal vessels. The injection of the loaded beads was performed as selective as possible using either a4F diagnostic catheter
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
Participants | 23 | 22

ADVERSE EVENTS:
Time Frame: 3 months
Description: Deterioration of liver functions Bleeding from puncture site Sepsis
Groups:
- Group 2: Twenty-five patients underwent conventional Chemoembolization (cTACE) using the standard TACE technique
  :TACE procedures were performed by experienced radiologists by fluoroscopy. The femoral artery was catheterized under local anesthesia, with a 4F catheter with Copra head configuration. Conventional angiography to delineate the feeding arteries of the tumors and to exclude portal venous shunting. Then vascular catheter was inserted super-selectively into the branch of the hepatic artery that is the main feeder of the tumor. Chemoembolization then was performed.
  Ten milliliters of Lipiodol was mixed with 100 mg of Doxorubicin hydrochloride and 5ml of Urografin emulsified to create a milky solution. The emulsion slowly was infused into the tumour Gel foam embolization was performedand an impirical antibiotic (gentamycin 80 mg). Injection of the mixture slowly under fluoroscopy guidance till complete stasis was achieved.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 1/25 | 5/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=25)
Deteriorating liver functions after the manouver (Hepatobiliary disorders) | 1 (1) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=25)
Bleeding from puncture site (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No